CLINICAL TRIAL: NCT00411281
Title: Treatment of Transient Myeloproliferative Disorder (TMD) in Children With Down Syndrome (DS)
Brief Title: Low-Dose Cytarabine in Treating Infants With Down Syndrome and Transient Myeloproliferative Disorder
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Per Group Chair: This study will not move forward.
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML0532; COG-AAML0532 (Other: Children's Oncology Group); CDR0000518352 (Other: Clinical Trials.gov)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2013-08

CONDITIONS: Leukemia
Keywords: acute myeloid leukemia/transient myeloproliferative disorder
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myeloproliferative Syndrome, Transient | interventions — Cytarabine; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Patients receive very low-dose cytarabine subcutaneously twice daily on days 1-7. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or complete or hepatic clinical remission undergo observation.
  Interventions: Drug: cytarabine
- Group II (Other): Patients are observed. If symptoms of intermediate- or high-risk disease develop, patients may crossover to group I.
  Interventions: Procedure: observation

INTERVENTIONS:
Drug: cytarabine — Given subcutaneously
  Arms: Group I
Procedure: observation — No intervention
  Arms: Group II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of abnormal cells, either by killing the cells or by stopping them from dividing. Giving low-doses of cytarabine may be an effective treatment for Down syndrome and transient myeloproliferative disorder. Sometimes the disease may not need treatment until it progresses. In this case, observation may be sufficient.

PURPOSE: This phase III trial is studying low-dose cytarabine to see how well it works in treating infants with Down syndrome and transient myeloproliferative disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether very low-dose cytarabine can improve event-free survival (EFS) rates in infants with high-risk transient myeloproliferative disorder (TMD), using high-risk TMD patients from clinical trial COG-A2971 for historic comparison, and in infants with intermediate-risk TMD, using intermediate-risk TMD patients from clinical trial COG-A2971 for historic comparison.
* Maintain the current high overall EFS rate in low-risk TMD patients.

Secondary

* Assess the toxicity of this regimen in these patients.

OUTLINE: This is a nonrandomized, multicenter, crossover study. Patients are stratified according to disease risk (high or intermediate vs low).

* Group I (patients with high- or intermediate-risk transient myeloproliferative disorder [TMD]): Patients receive very low-dose cytarabine subcutaneously twice daily on days 1-7. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or complete or hepatic clinical remission undergo observation.
* Group II (patients with low-risk TMD): Patients are observed. If symptoms of intermediate- or high-risk disease develop, patients may crossover to group I.

After completion of study treatment, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of transient myeloproliferative disorder (TMD)
* Diagnosis of Down syndrome or Down syndrome mosaicism (confirmed by karyotype analysis within the past 3 weeks) AND 1 of the following:

  * Nonerythroid and nonlymphoid blasts (any amount) in the peripheral blood with verification of a second sample
  * Trisomy 21-positive leukemic blasts documented by biopsy of any organ (including > 5% nonerythroid/nonlymphoid blasts documented by bone marrow aspirate or biopsy)
* Immunophenotype characterization required
* High-, intermediate-, or low-risk TMD, as defined by the following:

  * High-risk TMD, meeting 1 of the following criteria:

    * Life-threatening cardio-respiratory compromise due to complications of TMD (e.g., organomegaly or effusions)

      * Life-threatening cardio-respiratory compromise is defined as cardiovascular grade 4 edema, grade 4 pericardial effusions, or grade 4 pleural effusions
    * Hyperleukocytosis, defined as a WBC > 100,000/mm³
    * Any degree of hepatomegaly (palpable on physical exam) combined with life-threatening hepatic dysfunction

      * Life-threatening hepatic dysfunction is defined as grade 4 disseminated intravascular coagulation, grade 4 ascites, grade 4 bilirubin (> 10.0 times upper limit of normal [ULN]), or grade 4 AST or ALT (> 20.0 times ULN)
  * Intermediate-risk TMD, meeting all of the following criteria:

    * Hepatomegaly (palpable on physical exam) combined with non life-threatening hepatic dysfunction (i.e., grade 1-3 hepatic dysfunction [AST or ALT ≤ 2.5 times ULN] and/or a total or direct bilirubin ≤ 1.5 times ULN)
    * No evidence of life-threatening cardiovascular, respiratory, or hepatic compromise due to complications of TMD
  * Low-risk TMD, meeting all of the following criteria:

    * No palpable hepatomegaly on physical exam OR hepatomegaly is present without hepatic dysfunction (i.e., grade 0 hepatic dysfunction)
    * No evidence of life-threatening cardiovascular, respiratory, or hepatic compromise due to complications of TMD

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* No biliary atresia by hepatic ultrasound for patients with bilirubin 3.0-10.0 times ULN

PRIOR CONCURRENT THERAPY:

* No prior antileukemic therapy (except for leukapheresis or exchange transfusion)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Overall survival
Disease-related mortality
Percentage of patients experiencing grade 3-4 toxicity
Incidence of subsequent leukemia in patients for whom transient myeloproliferative disorder is resolved

CONTACTS AND LOCATIONS:
Overall Officials: April D. Sorrell, MD, Study Chair — Rutgers Cancer Institute of New Jersey; Jeffrey Taub, MD, Study Chair — Children's Hospital of Michigan